CLINICAL TRIAL: NCT00003079
Title: Phase I Study of Bryostatin 1 (NSC 339555) and High-Dose 1-Beta-D-Arabinofuranosylcytosine (HiDAC) in Patients With Refractory Leukemia
Brief Title: Bryostatin 1 and High Dose Cytarabine in Treating Patients With Refractory or Relapsed Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: National Cancer Institute
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065773; P30CA016059 (NIH); MCV-MCC-9612-2E; NCI-T97-0011
Record Dates: First submitted 2000-05-02; First posted 2004-05-27 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; recurrent adult lymphoblastic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — bryostatin 1; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bryostatin 1
Drug: cytarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of bryostatin 1 and high dose cytarabine in treating patients with refractory or relapsed acute myelocytic or acute lymphocytic leukemia, chronic myelogenous leukemia or refractory or relapsed lymphoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the maximum tolerated dose (MTD) of bryostatin 1 administered before and after high dose cytarabine in patients with refractory or relapsed acute myelocytic leukemia or acute lymphocytic leukemia, chronic myelogenous leukemia, or refractory or relapsed lymphoblastic lymphoma. II. Describe the toxic effects of bryostatin 1 and high dose cytarabine in these patients. III. Describe the time course of bryostatin 1 induced modulation of leukemic blast total protein kinase C (PKC) activity. IV. Describe bryostatin 1 pharmacokinetics. V. Correlate bryostatin 1 induced modulation of leukemic cell PKC activity or leukemic cell maturation with high dose cytarabine mediated apoptosis.

OUTLINE: This is a dose escalation study. Patients receive bryostatin 1 by continuous infusion over 24 hours on day 1. One hour after completion of bryostatin 1, patients receive high dose cytarabine IV over 3 hours every 12 hours on days 2-4. Patients again receive cytarabine over 3 hours every 12 hours on days 9-11, followed 1 hour later by bryostatin 1 by continuous infusion over 24 hours beginning on day 11. Patients achieving complete remission may receive up to 4 courses of consolidation chemotherapy. Consolidation chemotherapy is the same as induction chemotherapy except patients receive only 2 doses of cytarabine after day 1 completion of bryostatin and only 2 doses of cytarabine prior to the day 11 dose of bryostatin. Patients achieving partial remission may receive a second course of induction chemotherapy. In the absence of dose limiting toxicity in the first 3 patients treated, subsequent cohorts of 6 patients receive escalating doses of bryostatin 1 on the same schedule. If dose limiting toxicity occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the current dose is defined as the maximum tolerated dose. Patients are followed every 6 months until death.

PROJECTED ACCRUAL: A total of 12-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary refractory or relapsed acute myelocytic leukemia (AML) or acute lymphocytic leukemia (ALL), chronic myelogenous leukemia (CML) in blast crisis, or refractory or relapsed lymphoblastic lymphoma Priority is given to patients previously treated with conventional high dose cytarabine regimen without bryostatin 1 Eligible if previously failed a conventional high dose cytarabine regimen or if underwent subsequent high dose therapy with bone marrow/stem cell transplantation with curative intent

PATIENT CHARACTERISTICS: Age: 18 and over (must be 60 or under if receiving higher dose of cytarabine) Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL (bilirubin no greater than 3.0 mg/dL and conjugated bilirubin no greater than 0.5 mg/dL if Gilbert's disease and predominantly unconjugated hyperbilirubinemia present) AST no greater than 2.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine clearance at least 40 mL/min (at least 60 mL/min if receiving higher dose of cytarabine) Pulmonary: No clinically significant pulmonary disease Other: Not pregnant No patients who are poor medical risks because of nonmalignant systemic disease No serious, active, uncontrolled infection No prior or concurrent medical status that would make assessing cortical or cerebellar neurologic toxicity difficult

PRIOR CONCURRENT THERAPY: Recovery from the major toxic effects of prior therapy required Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 24 hours since prior chemotherapy with hydroxyurea At least 3 weeks since other prior systemic chemotherapy No prior clinically significant cerebellar toxicity due to cytarabine Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1997-09; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, MD, Study Chair — Massey Cancer Center
Locations (3):
- United States (3):
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center, Richmond, Virginia